CLINICAL TRIAL: NCT02702479
Title: Effect of Sucrose Versus High Fructose Corn Syrup on Cardiometabolic Risk: A Series of Systematic Reviews and Meta-Analyses of Controlled Trials
Brief Title: Meta-analyses of the Effect of Sucrose Versus High Fructose Corn Syrup on Cardiometabolic Risk
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Physicians' Services Incorporated Foundation (Other); Banting & Best Diabetes Centre (Other)
Responsible Party: Principal Investigator, John Sievenpiper, Associate Professor, University of Toronto
Other Study IDs: CIHR-Surose vs HFCS
Record Dates: First submitted 2016-03-02; First posted 2016-03-08 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Obesity; Dyslipidemia; Prediabetes; Dysglycemia; Gout; Hypertension; Non-Alcoholic Fatty Liver Disease; Cardiovascular Disease
Keywords: Systematic review and meta-analysis; Evidence-based medicine (EBM); Evidence-based nutrition (EBN); Clinical practice guidelines; Clinical trials; Dietary sugars; Fructose; High fructose corn syrup; Isocaloric; Hypercaloric; Cardiometabolic Risk Factors; Triglycerides; Cholesterol; Glycemic control; Body weight; Uric acid; Blood pressure; Fatty liver; Fasting; Postprandial
MeSH Terms: conditions — Obesity; Dyslipidemias; Prediabetic State; Gout; Hypertension; Non-alcoholic Fatty Liver Disease; Cardiovascular Diseases; Body Weight; Fatty Liver; Fasting | interventions — High Fructose Corn Syrup; Sucrose; Sugars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: High Fructose Corn Syrup — An intervention in which calories from HFCS are substituted isocalorically for sucrose in the diet
  Other Names: HFCS
Other: Sucrose — An intervention in which calories from sucrose are substituted isocalorically for HFCS in the diet
  Other Names: sugar

SUMMARY:
The rise in high fructose corn syrup (HFCS) consumption over the past 40 years since its introduction as a popular sweetener in the United States has led to much concern regarding its contribution to the rise in obesity (1), diabetes (2) and related cardiometabolic disorders (3).Unlike sucrose which contains equal proportions of fructose and glucose bound by an α-glycosidic bond, HFCS contains 42-55% of fructose to glucose in a free (unbound) form (4). Despite these differences in composition, both sugars possess identical energy contribution on a gram to gram basis (4). However, the higher ratio of fructose to glucose in HFCS has led to the hypothesis that HFCS may uniquely contribute to cardiometabolic risk, more so than sucrose, through proposed differences in fructose metabolism, endocrine and hedonic properties (5). We will conduct a series of systematic reviews and meta-analyses to assess the role of HFCS versus sucrose under energy matched (isocaloric) conditions on cardiometabolic risk.

DETAILED DESCRIPTION:
Need for proposed research: High quality systematic reviews and meta-analyses of controlled trials represent the highest level of evidence to support dietary guidelines and public health policy development. As HFCS has gained increasing popularity as a popular sweetener over the past ~50 years, replacing sucrose in the diet, there is an urgent need for systematic reviews and meta-analyses comparing sucrose versus HFCS in the development of cardiometaboilc diseases.

Objective: The investigators will conduct a series systematic reviews and meta-analyses to distinguish the effect of isocaloric exchange of sucrose versus HFCS on cardiometabolic risk in controlled trials.

Design: Each systematic review and meta-analysis will be conducted according to the Cochrane Handbook for Systematic Reviews of Interventions and reported according to the Preferred Reporting Items for Systematic Reviews and Meta-Analyses (PRISMA).

Data sources: MEDLINE, EMBASE, and The Cochrane Central Register of Controlled Trials (Clinical Trials; CENTRAL) will be searched using appropriate search terms supplemented by hand searches of references of included studies.

Study selection: The investigators will include randomized and non-randomized controlled trials >= 7-days in duration to assess the effect of sucrose versus HFCS under isocaloric conditions on measures of cardiometabolic risk. Direct comparisons of sucrose versus HFCS and indirect comparisons of sucrose or HFCS versus other carbohydrates under energy-matched conditions will be conducted.

Data extraction: Two or more investigators will independently extract relevant data and assess risk of bias using the Cochrane Risk of Bias Tool. All disagreements will be resolved by consensus. Standard computations and imputations will be used to derive missing variance data.

Outcomes: Seven sets of outcomes will be assessed: (1) body weight and markers of adipsoity (2) glycemic control, (3) blood pressure, (4) blood lipids, (5) uric acid, (6) non-alcoholic fatty liver disease (NAFLD) and ectopic fat, (7) inflammation

Data synthesis: Mean differences will be pooled using the generic inverse variance method when data are available from more than 2 trials. Random-effects models will be used even in the absence of statistically significant between-study heterogeneity, as they yield more conservative summary effect estimates in the presence of residual heterogeneity. Fixed-effects models will only be used where there is <5 included studies. Paired analyses will be applied for crossover trials. Heterogeneity will be assessed by the Cochran Q statistic and quantified by the I2 statistic. To explore sources of heterogeneity, the investigators will conduct sensitivity analyses, in which each study is systematically removed. If there are >=10 studies per endpoint, then the investigators will also explore sources of heterogeneity by a priori subgroup analyses by age (children [=<18 years of age], adults), health status (metabolic syndrome criteria, diabetes, overweight/ obese, healthy), comparator type, fructose- containing sugar form (sucrose, HFCS, honey, fructose), dose (=<10% energy, >10% energy), baseline measurements, randomization, study design (parallel, crossover), energy balance (positive, neutral, negative), follow-up (=<8-weeks, >8-weeks), and risk of bias. Meta-regression analyses will assess the significance of categorical and continuous subgroups analyses. When >=10 studies are available, publication bias will be investigated by inspection of funnel plots and formal testing using the Egger's and Begg's tests. If publication bias is suspected, then the investigators will attempt to adjust for funnel plot asymmetry by imputing the missing study data using the Duval and Tweedie trim and fill method.

Evidence Assessment: The strength of the evidence for each outcome will be assessed using the Grading of Recommendations Assessment, Development and Evaluation (GRADE).

Knowledge translation plan: The results will be disseminated through interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Target audiences will include the public health and scientific communities with interest in nutrition, diabetes, obesity, and cardiovascular disease. Feedback will be incorporated and used to improve the public health message and key areas for future research will be defined. Applicant/Co-applicant Decision Makers will network among opinion leaders to increase awareness and participate directly as committee members in the development of future guidelines.

Significance: The proposed project will aid in knowledge translation related to the role of sucrose versus HFCS in the development of cardiometabolic diseases, strengthening the evidence-base for guidelines and improving health outcomes by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

ELIGIBILITY:
Inclusion Criteria:

* Trials in humans
* Oral fructose-containing sugars intervention
* Presence of an adequate comparator in isocaloric substitution
* Diet duration >=7 days
* Viable outcome data

Exclusion Criteria:

* Non-human trials
* Observational studies
* IV or parenteral fructose-containing sugars
* Lack of suitable comparator (i.e. a comparator arm not including sucrose or HFCS in isocaloric substitution)
* Diet duration <7 days
* No viable outcome data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All individuals, both children and adults, regardless of health status.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Body weight and measures of adiposity analysis | Up to 20 years
Glycemic control analysis | Up to 20 years
Blood Lipids analysis | Up to 20 years
Blood pressure analysis | Up to 20 years
Uric acid analysis | Up to 20 years
Non-Alcoholic Fatty Liver Disease (NAFLD) and ectopic fat Analysis | Up to 20 years
Inflammation analysis | Up to 20 years

CONTACTS AND LOCATIONS:
Overall Officials: John L Sievenpiper, MD,PhD,FRCPC, Principal Investigator — University of Toronto
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada